CLINICAL TRIAL: NCT02302391
Title: Pharmacokinetic Analysis of Midazolam and Fentanyl in Pediatric Patients With Long-term Analgosedation.
Acronym: Morpheus
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr.med. Dominique Singer, Head of Section Neonatology and Pediatric Intensive Care, University Medical Center Hamburg-Eppendorf, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: PV4546
Record Dates: First submitted 2014-11-24; First posted 2014-11-27 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Deep Sedation; Intensive Care Pediatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Midazolam/fentanyl: PK analysis: Pediatric intensive care patients under analgosedation with midazolam and fentanyl.
  Interventions: Other: PK analysis

INTERVENTIONS:
Other: PK analysis — Quantification of Serum Levels and subsequent pharmacokinetic (PK) modelling.

SUMMARY:
Pharmacokinetic monitoring of midazolam, it's active metabolite and fentanyl in pediatric patients with long-term analgosedation will be performed. Especially, the chronologic sequence of the quantified plasma levels during sedation and during wake-up as well as the correlation to dose and sedation depth will be focused.

DETAILED DESCRIPTION:
At pre-defined timepoints (see below) serum Levels of the above mentioned drugs and metabolites will be determined and pharmakokinetic (PK) modeling will be performed. PK data will be correlated to sedation depth, as assessed using a validated score.

Three Age Groups (infants, children and adolescents) will be evaluated considering the physiologic properties during pediatric development.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients between 28 days and 17 years of age
* mechanical ventilation more than 3 days
* analgosedation with midazolam and fentanyl

Exclusion Criteria:

* missing informed consent

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with long-term analgosedation at the Pediatric Intensive Care Unit of the University Medical Center Hamburg-Eppendorf.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Plasma levels of midazolam, 1'-Hydroxymidazolam and fentanyl and resulting pharmacokinetic parameters | Once daily during analgosedation [expected average of 10 days) and 0, 1, 2, and 4h after stopping of midazolam

SECONDARY OUTCOMES:
Duration of mechanical ventilation | Participants will be followed for the duration of mechanical ventilation, an expected average of 10 days
Sedation depth | Participants will be followed for the duration of mechanical ventilation, an expected average of 10 days
Length of stay at the intensive care unit (ICU) | Participants will be followed for the duration of stay at the ICU, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Singer, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Department of Pediatrics
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany